CLINICAL TRIAL: NCT02070029
Title: Acupuncture in Premenopausal Women With Hypoactive Sexual Desire Disorder: A Prospective Cohort
Brief Title: Acupuncture for Sexual Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Collaborators: TriHealth Medical Education Research Fund (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12053
Record Dates: First submitted 2014-01-26; First posted 2014-02-24 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-02

CONDITIONS: Hypoactive Sexual Desire Disorder (HSDD); Low Libido; Female Sexual Dysfunction (FSD)
Keywords: Female Sexual Dysfunction (FSD); Hypoactive Sexual Desire Disorder (HSDD); Low libido; Acupuncture
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Acupuncture (Experimental): Acupuncture Therapy
  - twice weekly sessions for 5 weeks: 1st session 60 minutes with remaining 9 session approximately 45 minutes each. Physical exam at 1st session includes evaluation of peripheral pulses, head, neck, throat/tongue. No pelvic exam required.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture Therapy - Initial Evaluation History including: chief complaint, diet, level of diaphoresis, water intake, digestive function, menstrual cycling, sleep habits, overall mood.
  Physical Exam: inspection of tongue and palpation of central and peripheral pulses.
  Chinese Diagnoses for Female Sexual Dysfunction: Kidney Yang Deficiency; Liver Qi Stagnation; Generalized Blood Deficiency; Spleen Yang Deficiency; Heart Fire
  - Subsequent Sessions 25 minute sessions, twice weekly, for 5 weeks = total 10 sessions Needle usage = 8-20, average 14 per session Typically placed on the scalp, lower abdomen, elbows and knees

SUMMARY:
Female Sexual Dysfunction (FSD) affects up to 43% of women in the United States and Hypoactive Sexual Desire Disorder (HSDD) is the most common form. There is no standardized treatment for this condition. We know that alternative therapies such as acupuncture have been beneficial to women suffering from urinary incontinence, chronic lower back pain, and migraines. We hypothesize that the quality of life for premenopausal women with hypoactive sexual desire disorder (HSDD) will improve with initiation of acupuncture therapy for a duration of 5-weeks. Validated questionnaires are administered at the time of enrollment and 1 week after the final acupuncture session as the method of analyzing our primary outcome.

DETAILED DESCRIPTION:
Each woman will receive experimental therapy with acupuncture twice a week for five weeks and complete a packet of validated questionnaires/surveys at the 1st visit in person and at week 6 by mail.

The acupuncture sessions include:

* An Initial Evaluation in which the certified acupuncturist will take a
* History including: chief complaint, diet, level of diaphoresis, water intake, digestive function, menstrual cycling, sleep habits, overall mood
* Physical Exam: inspection of tongue and palpation of pulse
* 25 minutes of resting quietly with acupuncture needles in place
* Needle usage: from8 to 20 needles are typically used, with an average of 14 per session
* Needles are typically placed on the scalp, lower abdomen, elbows and knees

Subsequent Sessions (9 more) with the certified acupuncturist

* 25 minute each, twice weekly, for 5 weeks = total 10 sessions
* Needle usage = 8-20, average 14 per session
* Typically placed on the scalp, lower abdomen, elbows and knees

The questionnaires/surveys include questions about:

* Sexual desire, arousal, lubrication, orgasm, satisfaction and pain
* General physical health
* General emotional and psychological health
* Social relationships

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-55 years
* Sexually Active
* Premenopausal
* Documented diagnosis of HSDD as primary cause of FSD (defined as a non adjusted score of ≤ 6 in the desire domain of the FSFI questionnaire)

Exclusion Criteria:

* Postmenopausal, defined as absence of menstruation in the prior 12 months
* Pain or dyspareunia as the primary cause of FSD (defined as a non adjusted score of ≤ 6 in the pain domain of the FSFI)
* History of hysterectomy and/or oophorectomy
* History of chemotherapy, or pelvic irradiation
* Use of hormonal contraception or oral hormone replacement therapy
* Active skin infection or disease
* Blood dyscrasia
* Allergy to acupuncture needles

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Female Sexual Function Index (FSFI) | 6 weeks
  Determined by a change in the desire domain of the Female Sexual Function Index (FSFI) from baseline at enrollment to study completion at 6 weeks after initiation of intervention.

SECONDARY OUTCOMES:
Female Sexual Distress Scale (FSDS-R) | 6 weeks
  Determined by functional data points distributed at enrollment and 6 weeks:
  Female Sexual Distress scale - revised (FSDS-R)
Short Form-12 (SF-12) | 6 weeks
  Determined by functional data points distributed at enrollment and 6 weeks:
  Short Form-12 (SF-12)
Generalized Anxiety-Disorder-7 (GAD-7) and Prime Health Questionnaire-9 (PHQ-9) | 6 weeks
  Determined by functional data points distributed at enrollment and 6 weeks:
  Generalized Anxiety-Disorder-7 (GAD-7) and Prime Health Questionnaire-9 (PHQ-9)
World Health Organization Quality of Life- BREF (WHOQOL) | 6 weeks
  Determined by functional data points distributed at enrollment and 6 weeks:
  World Health Organization Quality of Life- BREF (WHOQOL)
Patient Global Impression of Improvement (PGI-I) | 6 weeks
  Determined by functional data points distributed at enrollment and 6 weeks:
  Patient Global Impression of Improvement (PGI-I)

CONTACTS AND LOCATIONS:
Locations (1):
- TriHealth, Cincinnati, Ohio, United States